CLINICAL TRIAL: NCT07393308
Title: Enhancing the Optimization of Empirical Antibiotic Therapy: Development and Implementation of Mobile Antibiograms in Tertiary Hospitals in Tanzania
Brief Title: Development and Implementation of Mobile Antibiograms to Optimize Empirical Antibiotic Prescriptions Among Prescribers in Tertiary Hospitals in Tanzania
Acronym: AMR; AMU; DDD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MUHAS-REC-10-2025-3152; 224127 (Other Grant/Funding Number: GSK Africa Open Lab)
Record Dates: First submitted 2026-01-21; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Antimicrobial Prescribing Practices; Antimicrobial Resistance (AMR)
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard of care (Active Comparator): Participants will be subjected to manual antibiogram which is the standard of care to guide the empirical prescription of antibiotics
  Interventions: Other: standard of care
- Mobile antibiogram (Experimental): Participants will be assigned to the mobile antibiogram application to guide the empirical prescription of antibiotics in addition to standard of care.
  Interventions: Other: Mobile antibiogram application

INTERVENTIONS:
Other: Mobile antibiogram application — A mobile antibiogram application software containing antibiotic sensitivity test results specific to the health facility. This mobile antibiogram application will guide decision support for empirical prescription.
  Arms: Mobile antibiogram
Other: standard of care — Participants will be assigned to manual antibiogram only.
  Arms: standard of care

SUMMARY:
Antimicrobial resistance (AMR) is a critical issue, especially in Africa, with resistance to common antibiotics reaching 100% in some areas. In Tanzania, limited access to culture tests and antibiograms forces healthcare providers to rely on experience for prescribing, heightening AMR risks. This study aims to determine the effectiveness of mobile antibiograms in optimizing empirical antibiotic therapy in tertiary hospitals in Tanzania.

DETAILED DESCRIPTION:
A pragmatic quasi-experimental design (hybrid type 1 trial) will be used to evaluate the effectiveness of mobile antibiograms on antibiotic use. The key role of the antibiogram is to guide empirical treatment of symptomatic infections using antibiotics ie., the antibiogram contains a list of susceptible and resistant antibiotics enabling the prescriber to rationally choose the antibiotic which is effective in clearing the infection. The study employs a three-phase, stepwise approach to assess and enhance antimicrobial use in Tanzanian hospitals. The first phase will be a baseline assessment using World Health Organization's Point Prevalence Survey and defined daily dose (DDD) to determine the pattern of antibiotic utilization and consumption respectively. The second phase involves developing a mobile antibiogram application through a participatory design with healthcare stakeholders. The final phase will use a quasi-experimental design to test the effectiveness of the mobile antibiogram on antimicrobial stewardship metrics like DDD per 1000 patient days, antibiotic appropriateness, infection-related mortality and length of hospital stay. The study sites will be Mbeya Zonal Referral Hospital (MZRH) as the intervention group and Benjamini Mkapa Hospital (BMH) as the control group. Additionally, a mixed-methods design (explanatory sequential design) will be used to assess the acceptability, feasibility, and adoption of the mobile antibiograms.

ELIGIBILITY:
Inclusion criteria

1. All prescribers working in the selected tertiary referral hospitals
2. All prescribers owning smartphones
3. Prescribers who consent to take part in the study

Exclusion criteria

1. Temporarily employed prescribers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Pattern of antibiotic use | 12 months
  Proportional change in antibiotic use among admitted patients

SECONDARY OUTCOMES:
Pattern of antibiotic resistance | 12 months
  Number of resistances to antibiotics among admitted patients
Acceptability of mobile antibiograms | 12 months
  % of acceptability of mobile antibiograms among prescribers
Feasibility of mobile antibiograms | 12 months
  % of feasibility mobile antibiogram among prescribers in tertiary referral hospitals in Tanzania
Adoption of mobile antibiogram | 12 months
  % of adoption of mobile antibiogram among prescribers in tertiary referral hospitals in Tanzania

CONTACTS AND LOCATIONS:
Locations (2):
- Tanzania (2):
  - Benjamin Mkapa Hospital, Dodoma
  - Mbeya Zonal Referral Hospital, Mbeya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zimbwe KB, Yona YJ, Chiwambo CA, Chandika AB, Kiwelu HS, Shabani MM. Trends and patterns of antimicrobial consumption at Benjamin Mkapa Zonal Referral Hospital, Dodoma, Tanzania: a cross-sectional retrospective analysis. BMJ Open. 2024 Nov 13;14(11):e083842. doi: 10.1136/bmjopen-2023-083842. PMID 39537568
- [Result] Shinohara KI, Yasuda S, Kato G, Fujita M, Shigekawa H. Direct measurement of the chiral quaternary structure in a pi-conjugated polymer at room temperature. J Am Chem Soc. 2001 Apr 18;123(15):3619-20. doi: 10.1021/ja003023m. No abstract available. PMID 11472144
- [Result] Mutagonda RF, Marealle AI, Nkinda L, Kibwana U, Maganda BA, Njiro BJ, Ndumwa HP, Kilonzi M, Mikomangwa WP, Mlyuka HJ, Felix FF, Myemba DT, Mwakawanga DL, Sambayi G, Kunambi PP, Ndayishimiye P, Sirili N, Mfaume R, Nshau A, Nyankesha E, Scherpbier R, Bwire GM. Determinants of misuse of antibiotics among parents of children attending clinics in regional referral hospitals in Tanzania. Sci Rep. 2022 Mar 22;12(1):4836. doi: 10.1038/s41598-022-08895-6. PMID 35318386
- [Result] Minzi OM, Kilonzi M, Mikomangwa WP, Bwire GM, Myemba DT, Marealle AI, Mlyuka HJ, Kibanga W, Mutagonda RF, Mwambete K. Update on bacterial and antibiotic susceptibility profiles among patients attending a tertiary referral hospital in Tanzania. J Glob Antimicrob Resist. 2021 Jun;25:87-88. doi: 10.1016/j.jgar.2021.02.030. Epub 2021 Mar 13. No abstract available. PMID 33727206
- [Result] Nkinda L, Mwakawanga DL, Kibwana UO, Mikomangwa WP, Myemba DT, Sirili N, Mwakalukwa R, Kilonzi M, Sambayi G, Maganda BA, Njiro BJ, Ndumwa HP, Mutagonda R, Marealle AI, Felix FF, Mlyuka HJ, Makuka G, Kubigwa SW, Kunambi PP, Mfaume R, Nshau AB, Bwire GM, Scherpbier R, Nyankesha E. Implementation of antibiotic stewardship programmes in paediatric patients in regional referral hospitals in Tanzania: experience from prescribers and dispensers. JAC Antimicrob Resist. 2022 Nov 23;4(6):dlac118. doi: 10.1093/jacamr/dlac118. eCollection 2022 Dec. PMID 36439992
- [Result] Costa-Paz M, Muscolo DL, Ayerza M, Makino A, Aponte-Tinao L. Magnetic resonance imaging follow-up study of bone bruises associated with anterior cruciate ligament ruptures. Arthroscopy. 2001 May;17(5):445-9. doi: 10.1053/jars.2001.23581. PMID 11337710
- [Result] Guerrier C, Wartanian R, Boblet V, Rohmer E, Le Lirzin R. [Cervical pregnancy. Contribution of ultrasonography to diagnosis and therapeutic management]. Rev Fr Gynecol Obstet. 1995 Jul-Sep;90(7-9):352, 355-9. French. PMID 7481440
- [Result] Fukunaga M, Tanaka C, Umeda M, Ebisu T, Aoki I, Watanabe Y, Higuchi T, Naruse S. Comparison of supplementary motor area activation between simple and complex motor task. Electroencephalogr Clin Neurophysiol Suppl. 1996;47:265-9. No abstract available. PMID 9335991
- [Result] Dorward AJ, Stack BH. Diffuse malignant pleural mesothelioma in Glasgow. Br J Dis Chest. 1981 Oct;75(4):397-402. doi: 10.1016/0007-0971(81)90027-9. PMID 7306467